CLINICAL TRIAL: NCT06627387
Title: A Low-Cost Balance Training Platform Using Augmented Reality in Neurorehabilitation: a Usability Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Eodyne Systems SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR(AT)309/2024
Record Dates: First submitted 2024-08-20; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Postural Balance; Cerebrovascular Disorders; Neurodegenerative Diseases; Augmented Reality; Neurological Rehabilitation
Keywords: Augmented Reality; Postural balance; Neurological Rehabilitation
MeSH Terms: conditions — Cerebrovascular Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: usability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Balance training (Experimental): The intervention will be carried out in two phases. The first phase will take place at Vall d'Hebron Hospital, where patients will undergo balance training under the supervision of a physiotherapist. The scheduled dose will be 60 minutes a day, 3 days a week for 4 weeks. If the patients meet the inclusion criteria, the intervention will be extended for two more weeks at home.
  Interventions: Other: Balance Training Using Augmented Reality

INTERVENTIONS:
Other: Balance Training Using Augmented Reality — The intervention will be carried out in two phases. The first phase will take place at Vall d'Hebron Hospital, where patients will undergo balance training under the supervision of a physiotherapist. The scheduled dose will be 60 minutes daily, three days a week for four weeks. If the patients meet the inclusion criteria, the intervention will be extended for two more weeks at home. For this task, the involvement of a family member as a training partner will be essential. Relatives will receive training on using the system in the hospital and must be present whenever the patient undergoes the training at home. Three assessments will be carried out during the six weeks of the study. At the beginning of the intervention ("Day 0" ), a second is once the hospital intervention has been carried out ("Week 4" ), and the last is once the home intervention has been carried out ("Week 6").
  Other Names: Personalized Health Assistance SystEM (PHASE)

SUMMARY:
The goal of this clinical trial is to assess the Usability, adherence, acceptance, and security of an augmented reality platform for balance training in patients with balance disorders due to degenerative injuries or cerebrovascular diseases.

The main questions it aims to answer are:

* Is the augmented reality system usable, acceptable, and safe with good adherence?
* Does the system improve the balance in our population?
* Participants will be asked to assist at Vall d'Hebrón Hospital, where patients will undergo balance training under the supervision of a physiotherapist three days a week for four weeks.
* If the patients meet the inclusion criteria, the intervention will be extended for two more weeks at home.

DETAILED DESCRIPTION:
2. INTERVENTION The first phase of the intervention will last four weeks and will be done in the hospital. After this intervention, if the patients meet the inclusion criteria, they will be enrolled in the second phase, which will be done at the patient's home for two additional weeks. Three assessments will be performed during the study: The first one ("Day 0") will be assessed before starting the treatment, the second one will be done ("Week 4") directly after the intervention at a hospital setting, and the last one ("Week 6"), after the home intervention. The intervention will be conducted in 1-hour sessions three times a week for four weeks, performing different exercises using an augmented reality platform accessed through RGSweb. If the patients continue the intervention at home, a three-session training for two weeks will be conducted in the presence of a patient's relative, who will accept to be the training partner.

3. EQUIPMENT AND TECHNICAL SPECIFICATIONS. RGSweb can be used with any computer or device with a camera. However, our target users are patients who might have visibility issues due to old age. Therefore, bigger screens will be used to enhance the patients'; visibility. Additional screen support will be required to hold the monitor.

There are three protocols in RGSweb:

Twister Buddy: It has been developed for balance training, which involves a series of levels intended to strengthen the muscles crucial for maintaining upright posture, notably those in the legs. The aim is to improve stability and help prevent falls.

Levels The user will have to shift their weight from one leg to the other while doing different exercises, such as touching targets with their hands and feet or taking steps.

All levels will start with a calibration phase to ensure the user is in the correct position.

Level 1 -Balance: In this level, two colored columns will be displayed on the screen, while user motion trackers will also be reflected on the screen. The goal is to align the trackers with the same color column.

Level 2 - Balance + Hands: In addition to the balance movement from Level 1, a target will be displayed on the screen. The user must maintain balance on the highlighted column while reaching the target with their hand.

Level 3 - Side Steps: To initiate, the user must have their feet on a square-like target at the bottom center of the screen. After that, a target will appear adjacent to the square. The user's task is to adjust their foot position so that both the toe and heel are inside this target area. Once achieved, the user must return their foot to the original position within the square, prompting the appearance of the next target for the opposite foot.

Level 4 - Front steps: Similar to level 4, the user begins by positioning both feet on the square target. Then, an arrow will appear above one of the user's feet, indicating the direction of the step (either forward or backward). Once the user moves the designated foot past a predefined threshold value, currently indicated by a slider, the arrow will disappear, prompting the user to return both feet to the square. Subsequently, an arrow will appear above the other foot, indicating the direction for the next step. The direction of the steps is randomized for each interaction.

Level 5 -- Balance + Hands + Feet: This is the next step from level 4. It starts with Balance, then the target for the hand, and finally, the target for the opposite foot. Like level 2, the user must maintain only the bottom part (hip and under) inside the column while reaching the target with their hand and foot.

Costume Party: This protocol's main focus is sit-to-stand. The levels of this exercise follow different steps to stand up from a chair, starting with leaning forward.

Levels All levels will start with a calibration phase to ensure the user is in the correct position.

The objective is to dress up for a costume party using a reference shown at the bottom right of the screen. Various costume parts will appear on a bar and move across the screen. The user needs to catch the right parts for their costume and put them on. Once the costume is complete, there will be a few seconds to admire it before the process starts over with a new costume reference.

Level 1-Lean Forward: In this level, the costume elements move from one side of the screen to another at the user's eye level.

To grab the element, they must lean forward enough to surpass a threshold value defined by a slider.

Level 2-Flex Knees: The user starts the motion of standing up by flexing the knees and rising slightly from the chair.

The elements will appear close to the user's head, and leaning forward is unnecessary.

Level 3-Stand Up: This level is similar to level 2, but the elements are positioned higher, requiring the user to stand up to reach them.

Gentle Giant: This exercise targets less-impaired patients who can perform sit-to-stand and balance training exercises.

Levels:

The aim is to allow the elements to move from one platform to another following color coding. To do so, the user will act as a bridge between the different floors.

All levels will start with a calibration phase to ensure the user is in the correct position.

Level 1-Squats: In this level, the user must move the elements from one platform to another by moving the bridge up and down, that is, by squatting to go down and standing again to come up.

Level 2-Tip-Toe: In this level, one platform will be higher than the user's height. The aim is similar, though: The user must stand in a tip-toe position to move the bridge higher and connect the platforms.

ELIGIBILITY:
Inclusion Criteria:

* Balance impairment due cerebrovascular diseases or neurodegenerative diseases.
* Being able to mantain standing for 2 minuts without assistance.
* Berg scale ≥21
* Age ≥18
* Signing informed consent
* To have a training partner during the exercises at home.
* No fall attempt during hospital intervention
* No have enough space to train safely at their home.
* Being familiar with technological devices such a laptop, tablets or inteligent cellphones.

Exclusion Criteria:

* The presence of a condition or abnormality that could compromise the patient's safety.
* Severe cognitive impairments tha prevent the execution of the xperiment (MoCA <19)
* Presence of sensory aphasia.
* Diagnostic of conduct disorders.
* Presence of severe neglect.
* Spasticity =4 in MAS lower limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | "Week 4" "Week 6"
  The System Usability Scale is a reliable tool for measuring usability. It consists of a 10-item questionnaire with five response options for respondents, from Strongly Agree to Disagree Strongly. A value above 68 points is considered acceptable.
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) | "Week 4" "Week 6"
  The instrument is a self-administered questionnaire assessing user satisfaction with assistive technology product and associated services.
User Esperience Questionnaire (UEQ) | "Week 4" "Week 6"
  The scales of the questionnaire cover comprehensive impression of user experience. Both classical usability aspects (efficiency, perspicuity, dependability) and user experience (originality stimulation) are measured. The items are scaled from -3 to +3. Thus, -3 represents the most negative answer, 0 a neutral answer, and +3 the most positive answer.
Adherence (Home) | "Week 6"
  Time the Augmentad reality system is used in comparision to the scheduled dosage.
Adherence (Hospital) | "Week 4"
  Total sessions scheduled for therapy compared to the number of sessions attended
Ad-hoc questions | "Day 0" "Week 4" "Week 6"
  Questions to assess the attitude towards the system and to gather data on privacy and feeling of stigma.

SECONDARY OUTCOMES:
Berg Balance Scale | "Day 0" "Week 4" "Week 6"
  The Berg Balance Scale is a 14-item scale that assesses balance and fall risk in adults. Patients receive a score from 0-4 on their ability to meet these balance dimensions. A global score can be calculated out of 56. A score of 0 represents an inability to complete the item, and a score of 56 represents the ability to independently complete the item.
Postural Sway | "Day 0" "Week 4" "Week 6"
  Quantitative static balance assement. It will be assessed using Ned SVE/IBE system for postural assessment.
Five Times Sit to Stand Test (FTSS) | "Day 0" "Week 4" "Week 6"
  The Five Times Sit to Stand Test is a highly reliable tool for assessing lower limbs strengh and balance control and is used to detect risk of fall in enderly and stroke patients. In this test the participants are instructed to stand up from a chair five times as fast as possible.
The Activities-specific Balance Confidence (ABC) Scale. | "Day 0" "Week 4" "Week 6"
  &-item self-report measure in wich patients rate their balance confidence for performing activities.
The EuroQol-5 Dimension-5 Level (EQ-5D-5L) | "Day 0" "Week 4" "Week 6"
  It is a self-report survey that measures quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "No problems" to "Extreme problems."

OTHER OUTCOMES:
The Montreal Cognitive Assesment (MoCA) | "Day 0"
  Cognitive test validated as a highly sensitive tool for early detection of mild cognitive impairment. MoCA assesses short term memory, visuospacial abilities, executive functions, attention, concentration and working memory, and orientation to time and place.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Rodriguez Gonzalez, MD, Principal Investigator — VHIR
Locations (1):
- Hospital Vall D'Hebrón, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
We are the only center involved in the studdy and we don't consider to share patients data with other researchers.

REFERENCES:
- [Background] Truijen S, Abdullahi A, Bijsterbosch D, van Zoest E, Conijn M, Wang Y, Struyf N, Saeys W. Effect of home-based virtual reality training and telerehabilitation on balance in individuals with Parkinson disease, multiple sclerosis, and stroke: a systematic review and meta-analysis. Neurol Sci. 2022 May;43(5):2995-3006. doi: 10.1007/s10072-021-05855-2. Epub 2022 Feb 17. PMID 35175439
- [Background] Lim JH, Lee HS, Song CS. Home-based rehabilitation programs on postural balance, walking, and quality of life in patients with stroke: A single-blind, randomized controlled trial. Medicine (Baltimore). 2021 Sep 3;100(35):e27154. doi: 10.1097/MD.0000000000027154. PMID 34477171
- [Background] Keller JL, Bastian AJ. A home balance exercise program improves walking in people with cerebellar ataxia. Neurorehabil Neural Repair. 2014 Oct;28(8):770-8. doi: 10.1177/1545968314522350. Epub 2014 Feb 13. PMID 24526707
- [Background] Lei C, Sunzi K, Dai F, Liu X, Wang Y, Zhang B, He L, Ju M. Effects of virtual reality rehabilitation training on gait and balance in patients with Parkinson's disease: A systematic review. PLoS One. 2019 Nov 7;14(11):e0224819. doi: 10.1371/journal.pone.0224819. eCollection 2019. PMID 31697777
- [Background] Iruthayarajah J, McIntyre A, Cotoi A, Macaluso S, Teasell R. The use of virtual reality for balance among individuals with chronic stroke: a systematic review and meta-analysis. Top Stroke Rehabil. 2017 Jan;24(1):68-79. doi: 10.1080/10749357.2016.1192361. Epub 2016 Jun 16. PMID 27309680